CLINICAL TRIAL: NCT05027685
Title: The "Global Paradise® System" Registry
Brief Title: The "Global Paradise System" Registry
Acronym: GPS Registry
Status: Recruiting | Type: Observational
Sponsor: ReCor Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN-0927
Record Dates: First submitted 2021-07-26; First posted 2021-08-30 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Hypertension
Keywords: Hypertension; Blood pressure; Renal Denervation
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Renal Denervation Treatment: Patients candidate for treatment or already treated within 6 months prior to consent, as per the sites normal practice with the commercially available Paradise Ultrasound Renal Denervation System, will be enrolled in this single arm registry.
  Interventions: Device: The Paradise Ultrasound Renal Denervation System

INTERVENTIONS:
Device: The Paradise Ultrasound Renal Denervation System — The CE-marked and commercially available ReCor Medical Paradise Ultrasound Renal Denervation System (Paradise System) is a catheter-based device designed to use ultrasound energy to thermally ablate the nerves surrounding the renal artery and serving the kidney.

SUMMARY:
The GPS Registry is a multi-centre, single-arm, non-interventional (observational) registry. In addition to collecting data from patients treated as per standard clinical practice, the Registry will also regularly collect telemetric Home Blood Pressure (HBP) measurements and Patient Reported Outcome (PRO) data via a standardized quality of life questionnaire. The objective of the GPS Registry is to document the long-term safety and effectiveness of the commercially available Paradise Ultrasound Renal Denervation System when used per its labelling in patients deemed to be candidates for RDN as per physician's assessment.

ELIGIBILITY:
Inclusion Criteria:

* Appropriately signed and dated informed consent
* Age ≥18 at time of consent
* Patient candidate for renal denervation with the Paradise System based on physician's assessment OR Patient treated with the Paradise Ultrasound Renal Denervation System within the 6 months prior to consent

Exclusion Criteria:

Patients who meet any of the contraindications listed in the Instructions for Use will be excluded.

The contraindications are:

* Stented renal artery
* Less than 18 years of age
* Pregnant
* Known allergy to contrast medium
* Renal arteries diameter < 3 mm and > 8 mm
* Renal artery with Fibromuscular (FMD) disease
* Renal artery aneurysm
* Renal artery stenosis of any origin >30%
* Iliac/femoral artery stenosis precluding insertion of the Paradise catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The GPS Registry will collect both retrospective and prospective data in patients treated as per the sites normal practice with the commercially available Paradise Ultrasound Renal Denervation System.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-01-13 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of all-cause mortality | Through 5 Years post-procedure
  Rate of mortality attributed to any causality as per site standard practice.
Incidence of new onset end-stage renal disease | Through 5 Years post-procedure
  eGFR<15 mL/min/m2 or need for renal replacement therapy as per site standard practice
Significant decline in renal function | Through 5 Years post-procedure
  ≥50% increase in serum creatinine (mg/dL)
New renal artery stenosis | Through 5 Years post-procedure
  >70% confirmed by CTA/MRA as per site standard practice.
Incidence of renal artery perforation or dissection requiring an invasive intervention | Through 5 Years post-procedure
Incidence of major vascular complications (e.g, clinically significant groin hematoma, arteriovenous fistula, pseudoaneurysm) requiring surgical repair, interventional procedure, thrombin injection, or blood transfusion as per site standard practice | Through 5 Years post-procedure
Incidence of hospitalization for hypertensive crisis or symptomatic hypotension | Through 5 Years post-procedure
Incidence of hospitalization for major cardiovascular- or hemodynamic-related events (e.g. HF; AF) | Through 5 Years post-procedure
Incidence of new onset stroke, TIA or CVA | Through 5 Years post-procedure
Incidence of acute myocardial infarction | Through 5 Years post-procedure
Incidence of any coronary revascularization | Through 5 Years post-procedure
Reduction in average home systolic/diastolic BP in mmHg as compared to enrollment | Through 5 Years post-procedure
Reduction in average office systolic/diastolic BP in mmHg as compared to enrollment | Through 5 Years post-procedure
Reduction in average ambulatory systolic/diastolic BP in mmHg (daytime, nighttime and 24-hr) as compared to enrollment | Through 5 Years post-procedure
Incidence of home systolic BP reductions of ≥5 mmHg, ≥10 mmHg, and ≥15 mmHg | Through 5 Years post-procedure
Incidence of office systolic BP reductions of ≥5 mmHg, ≥10 mmHg, and ≥15 mmHg | Through 5 Years post-procedure
Incidence of ambulatory systolic BP (daytime/24-hr/night-time) reductions of ≥5 mmHg, ≥10 mmHg, and ≥15 mmHg | Through 5 Years post-procedure
Percentage of subjects who are controlled according to current guidelines | Through 5 Years post-procedure
Change in office/home/ambulatory pulse pressure in mmHg | Through 5 Years post-procedure
Change in office/home/ambulatory heart rate in bpm | Through 5 Years post-procedure
Percentage of subjects without any anti-hypertensive treatment with analysis stratified by number of enrollment antihypertensive medications | Through 5 Years post-procedure
Analysis of quarterly Home BP in mmHg | Through 5 Years post-procedure
Change from enrollment in quality of life scores as measured by the 12-item Short Form Health Survey (SF-12) | Through 5 Years post-procedure
  The 12-item Short Form Health Survey (SF-12) is a measure of health-related quality-of-life. Scores for each domain range from 0 to 100, with a higher score indicating a more favorable health state.

CONTACTS AND LOCATIONS:
Overall Officials: Melvin Lobo, Prof., Principal Investigator — Barts NIHR Biomedical Research Centre, William Harvey Research Institute, QMUL; Felix Mahfoud, Prof., Principal Investigator — UKS Universitätsklinikum des Saarlandes, Kardiologie, Angiologie und internistische Intensivmedizin
Locations (35):
- Belgium (3):
  - OLV Ziekenhuis Aalst, Aalst
  - CHU Saint Pierre Brussels, Brussels
  - UCL St Luc, Brussels
- France (3):
  - CHU Bordeaux Hôpital St. André, Bordeaux
  - HEGP (Hôpital Européen Georges Pompidouv) Paris, Paris
  - Centre Hospitalier de Pau, Pau
- Germany (17):
  - Universitäts-Herzzentrum Freiburg Bad Krozingen, Bad Krozingen
  - Charité Universitätsmedizin Berlin Campus Benjamin Franklin, Berlin
  - Klinikum Coburg GmbH, Coburg
  - Universitätsklinikum Köln, Cologne
  - Klinikum Lippe GmbH Detmold, Detmold
  - Herzzentrum Dresden GmbH Universitätsklinik, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Erlangen, Erlangen
  - Cardiovasculäres Centrum (CVC) Frankfurt, Frankfurt
  - St. Barbara-Klinik Hamm Heessen, Hamm
  - University Clinic of Saarland - Homburg, Homburg
  - Herzzentrum Leipzig GmbH, Leipzig
  - Sana Kliniken Lübeck gGmbH, Lübeck
  - Marienhaus Klinikum Mainz, Mainz
  - Detusches Herzzentrum München (DHM), München
  - Robert-Bosch-Krankenhaus GmbH Stuttgart, Stuttgart
  - Schwarzwald-Baar Klinikum Villingen-Schwenningen, Villingen-Schwenningen
- Centre Hospitalier Princesse Grace Monaco, Monaco, Monaco
- Netherlands (2):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Erasmus MC Rotterdam, Rotterdam
- Switzerland (2):
  - HUG Geneve Switzerland, Geneva
  - Heart Center Lucerne -Luzerner Kantonsspital, Lucerne
- United Kingdom (7):
  - Royal Bournemouth Hospital, Bournemoth, Bournemouth
  - Kent and Canterbury Hospital, Canterbury, Canterbury
  - University Hospital Wales, Cardiff, Cardiff
  - Queen Elizabeth Hospital, Glasgow, Glasgow
  - Hammersmith Hospital (Imperial College Healthcare NHS Trust), London
  - WHRC - Barts Health, London, London
  - Freeman Hospital, Newcastle, Newcastle